CLINICAL TRIAL: NCT04735029
Title: A Randomized Controlled Trial on the Effect of Focal Thermal Therapy at Acupuncture Points in the Treatment of Osteoarthritis of the Knee
Brief Title: Focal Thermal Therapy Acupoint OA Knee RCT
Acronym: ThermAcuRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ho Ki Wai, Clinical Professional Consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016.555-T
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis, Knee; Randomized Controlled Trial
Keywords: knee osteoarthritis; acupuncture; randomized control trial
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Group 1: Heat pack group; Group 2: Thermal Gun group
Who Masked: Participant, Care Provider
Masking Description: Envelope
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermal Gun group (Experimental): The thermal gun applied on acupressure points in TCM. The thermal gun used a heat-generating ceramic head to apply a dual effect called "heat-and-light-pressure" on the acupuncture points.
  Interventions: Device: Thermal gun
- Heat Pack group (Active Comparator): A hydrocollator heat pack used to simulate traditional thermal therapy. The application of the heat pack was wrapped with six layers of terry towels to bring the temperature down to around 43°C.
  Interventions: Other: Heat pack

INTERVENTIONS:
Device: Thermal gun — Thermal gun used a heat-generating ceramic head to apply a dual effect called "heat-and-light-pressure" on the acupuncture points.
  Arms: Thermal Gun group
Other: Heat pack — A hydrocollator heat pack used to simulate traditional thermal therapy
  Arms: Heat Pack group

SUMMARY:
Osteoarthritis of the knee is a common degenerative joint disorder in our ageing population. A combination of thermal therapy with a self-management exercise have shown a positive effect in the management of osteoarthritis of the knee. This study aimed to compare the effectiveness of topical heat pack versus focal application of heat therapy at the acupressure points in the treatment of osteoarthritis of the knee.

DETAILED DESCRIPTION:
Osteoarthritis of the knee is a common degenerative joint disorder in our ageing population. A combination of thermal therapy with a self-management exercise have shown a positive effect in the management of osteoarthritis of the knee. This study aimed to compare the effectiveness of topical heat pack versus focal application of heat therapy at the acupressure points in the treatment of osteoarthritis of the knee.

A randomized control trial was conducted in 76 patients with osteoarthritis of the knee, diagnosed by an experienced orthopedic surgeon. Following inclusion and exclusion selection, patients were randomly allocated to group 1 (Heat Pack) or group 2 (Thermal Gun). All patients received 30 minutes of treatment in each session, twice a week for 4 weeks. They also received an education program and taught home knee exercises. Outcome measurements were Visual Analog Scale (VAS) for pain intensity, muscle power, knee ROM, WOMAC and SF-12v2.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients aged 40 years old or older
* clinical and radiological diagnosis of osteoarthritis of the knee based on the OA Knee clinical guidelines and radiological evidence
* normal skin sensation to heat, cold, pins and pricks (i.e. passed the required Skin Sensation Test)
* not participating in any other clinical trial at time of this study
* be able to complete the whole trial period
* no cognitive dysfunction and was able to sign the consent form

Exclusion Criteria:

* received bilateral knee arthroplasty before this study
* polyarthritis affecting more than both knee
* active skin lesion
* women in pregnancy or breasts feeding
* received acupuncture and/or moxibustion within one month of the study
* unable to comply with the study protocol

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) for pain | Baseline
  10-scale likert scale to measure pain level visually; Minimum = 0 and Maximum value = 10, and higher scores mean a better outcome.
Visual analogue scale (VAS) for pain | After 1 year
  10-scale likert scale to measure pain level visually; Minimum = 0 and Maximum value = 10, and higher scores mean a better outcome.
Knee range of movement (ROM) | Baseline
  Knee range of movement (ROM) in the supine position using a goniometer; Numeric
Knee range of movement (ROM) | After 1 year
  Knee range of movement (ROM) in the supine position using a goniometer; Numeric
Quadriceps and hamstrings muscle strength | Baseline
  Quadriceps and hamstrings muscle strength were measured according to the Oxford Scale of Muscle Strength; Numeric
Quadriceps and hamstrings muscle strength | After 1 year
  Quadriceps and hamstrings muscle strength were measured according to the Oxford Scale of Muscle Strength; Numeric
Western Ontario and McMasters Universities (WOMAC) | Baseline
  Functional assessment with the validated Chinese version of the Western Ontario and McMasters Universities (WOMAC); Numeric
Western Ontario and McMasters Universities (WOMAC) | After 1 year
  Functional assessment with the validated Chinese version of the Western Ontario and McMasters Universities (WOMAC); Numeric
Short Form-12 version 2 (SF-12v2) | Baseline
  Quality of life evaluation; Expressed by Physical component summary (PCS) and Mental component summary (MCS); Both numeric, The higher score the better outcome
Short Form-12 version 2 (SF-12v2) | After 1 year
  Quality of life evaluation; Expressed by Physical component summary (PCS) and Mental component summary (MCS); Both numeric, The higher score the better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Ki-Wai Ho, Study Director — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho KK, Kwok AW, Chau WW, Xia SM, Wang YL, Cheng JC. A randomized controlled trial on the effect of focal thermal therapy at acupressure points treating osteoarthritis of the knee. J Orthop Surg Res. 2021 Apr 27;16(1):282. doi: 10.1186/s13018-021-02398-2. PMID 33906695